CLINICAL TRIAL: NCT00073086
Title: Clinical Evaluation and Management of Persons With Severe Acute Respiratory Syndrome (SARS)
Brief Title: Evaluation and Treatment of Severe Acute Respiratory Syndrome (SARS)
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040030; 04-I-0030
Record Dates: First submitted 2003-11-14; First posted 2003-11-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-27

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: Coronavirus; Pneumonia; Asia; China; Severe Acut Respiratory Syndrome; SARS; Suspected SARS
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections; Pneumonia

SUMMARY:
This study will evaluate and treat people with SARS, a new type of pneumonia (lung infection) originating in China. SARS is caused by a new virus that is easily transmitted from person to person. This study will look at the course of the disease; determine how the virus affects the body and how the body fights the infection; and evaluate diagnostic tests to quickly identify the disease.

People 18 years of age and older with probable or suspected SARS may be eligible for this study. Close contacts of patients with SARS, patients who recovered from SARS, and NIH health care workers involved in the care of patients will also be enrolled. Patients with SARS who require hospitalization will be admitted to the NIH Clinical Center. Because SARS spreads easily, hospitalized patients will be in a room by themselves and will not be allowed any visitors. They will not leave their room except for tests, such as x-rays.

All participants will have a full medical examination, including a medical history, physical examination, and blood tests. In addition, the participants undergo various tests and procedures as follows:

* Probable and suspected SARS patients may be hospitalized or may be seen as outpatients. They are provided the treatment judged best for their disease, usually according to expressed or published recommendations. The best treatment for SARS is not yet known, and there have been no studies evaluating therapies. Outpatients are seen three times a week for 2 weeks, once a week for 4 more weeks, and then at 6 months. Patients have mouth and throat swabs taken three times a week for the first 2 weeks, then once a week for 4 more weeks. Blood is drawn three times a week for the first 2 weeks, then once at weeks 3, 4, and 6. If virus is still detectable after 6 weeks, nose washings and throat swabs are repeated until no virus is detected for 3 weeks in a row. In addition, patients provide urine and stool samples, have a chest x-ray and electrocardiogram, and undergo bronchoscopy and bronchial lavage. For the bronchoscopy, a bronchoscope (pencil-thin flexible tube) is passed into the large airways of the lung, allowing the physician to examine the airways. Cells and secretions from the airways are rinsed from the lung with salt water. A brush the size of a pencil tip is passed through the bronchoscope to scrape cells lining the airways and pieces of tissue are collected for analysis.
* Close contacts of patients are evaluated twice a week for 2 weeks, then once a week for 2 more weeks. Blood is drawn at the first visit and then at 1, 2, and 4 weeks. Mouth and throat swabs, nose washings, and sputum collections are done twice a week for 2 weeks, then once a week for 2 more weeks. Urine and stool samples are collected once a week for 4 weeks. If virus from the nose or throat is still detectable after 4 weeks, weekly nose washings and throat swabs continue until no virus is detected for 3 weeks in a row. Blood may also be drawn during the weekly visits.
* Recovered SARS patients provide blood, urine, and stool samples and have a mouth and throat swab and nose aspiration to see if the SARS virus is present. For the nasal aspiration, salt water is put in the nose and then suctioned out. Usually, these tests are done only once. If virus is detected, however, the nose washing, throat swabs and blood tests are repeated once a week until no virus is detected for 3 weeks in a row.
* Health care workers document their contact with patients, use of isolation procedures and equipment, and any unexpected events that occur during contact. They are evaluated for symptoms of infection and provide a blood sample once a month

DETAILED DESCRIPTION:
Since mid February 2003, there have been reports of atypical pneumonias originating in China which have subsequently been termed the Severe Acute Respiratory Syndrome (SARS). SARS has subsequently spread to multiple countries including the United States, and is accompanied by a higher than anticipated morbidity and mortality. Because of world travel and the apparent easy transmissibility of this disease reported in other nations, the number of patients with SARS may continue to rise. The primary purpose of this protocol is to evaluate and treat persons with SARS. Other goals will be to characterize the clinical course of SARS by also evaluating close contacts of people with SARS, as well as those that have recovered from SARS. Additional goals of the protocol are to elucidate the pathophysiology of SARS, characterize the immune response during SARS, and evaluate diagnostic tests for the rapid identification of SARS in clinical specimens. Further knowledge about SARS may lead to effective forms of therapy and improve mortality from this disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Probable SARS Inclusion Criteria:

1. One of the following:

   Travel within 10 days of onset of symptoms to an area with documented or suspected community transmission of SARS (as continually defined by the WHO and/or CDC)

   OR

   Close contact within 10 days of onset of symptoms with a person known to be a suspect SARS case.

   Close contact is defined as having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient known to be suspect SARS case.

   AND
2. Measured temperature greater than 100.4(Degree)F (greater than 38(Degree) C)

   AND
3. Evidence of an acute respiratory illness as manifested by one of the following:

   Cough: shortness of breath, difficulty breathing, hypoxia

   AND
4. Radiographic evidence of pneumonia or ARDS

   AND
5. Clinically stable for transfer to the Clinical Center

   AND
6. The ability to understand and willingness to sign a written consent form or in cases of 1) a minor, 2) temporary incompetence due to severe illness, or 3) permanent incompetence due to a chronic condition, informed consent may be signed by a legal guardian or appropriate proxy.

Suspected SARS Inclusion Criteria:

1. One of the following:

   1. Travel within 14 days of onset of symptoms to an area with documented or suspected community transmission of SARS (as continually defined by the WHO and/or CDC)

      OR
   2. Close contact within 14 days of onset of symptoms with either a person with a respiratory illness who traveled to a SARS area or a person known to be a suspect SARS case.

   Close contact is defined as one of the following:

   Close contact is defined as having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient known to be suspect SARS case.

   Other contact of sufficient proximity and duration that transmission of the causative agent of SARS may have occurred. This will be determined on an individual basis by the PI or an associate investigator.

   AND
2. One of the following:

   1. Measured temperature greater than 100.4(Degree)F (greater than 38(Degree) C)
   2. Evidence of an acute respiratory illness as manifest by one of the following:

   cough, shortness of breath, difficulty breathing, hypoxia, radiographic findings of either pneumonia or acute respiratory distress syndrome

   AND
3. Clinically stable for transfer to the Clinical Center

   AND
4. The ability to understand and willingness to sign a written consent form or in cases of 1) a minor, 2) temporary incompetence due to severe illness, or 3) permanent incompetence due to a chronic condition, informed consent may be signed by a legal guardian or appropriate proxy.

Close Contact Inclusion Criteria:

1. Close contact with a patient suspected to have SARS within 10 days of the time of enrollment.

   Close contact is defined as one of the following:

   having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient suspected or known to have SARS.

   Other contact of sufficient proximity and duration that transmission of the causative agent of SARS may have occurred. This will be determined on an individual basis by the PI or an associate investigator.

   AND
2. The ability to understand and willingness to sign a written consent form or in cases of 1) a minor, 2) temporary incompetence due to severe illness, or 3) permanent incompetence due to a chronic condition, informed consent signed by a legal guardian or appropriate proxy.

Recovered SARS Inclusion Criteria

1. Within the last six months, had one of the following:

1. an acute illness characterized by (all of the following):

   1. Fever greater than 100.4 (if measured)

      AND
   2. History of an acute respiratory illness as manifested by one of the following:

      cough, shortness of breath, difficulty breathing, hypoxia

      AND
   3. The illness occurred within 10days of travel to an area with documented or suspected community transmission of SARS (as continually defined by the WHO and/or CDC)

   OR

   Had close contact within 10 days of onset of symptoms with either a person with a respiratory illness who traveled to a SARS area or a person known to be a suspected SARS case.

   Close contact is defined as one of the following:

   Close contact is defined as having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient known to be suspect SARS case.

   Other contact of sufficient proximity and duration that transmission of the causative agent of SARS may have occurred. This will be determined on an individual basis by the PI or an associate investigator.

   OR
2. an acute respiratory illness with the laboratory confirmation of SARS

   AND

   2. The ability to understand and willingness to sign a written consent form or in cases of 1) a minor, 2) temporary incompetence due to severe illness, or 3) permanent incompetence due to a chronic condition, informed consent signed by a legal guardian or appropriate proxy.

   Health Care Worker Surveillance Inclusion Criteria
   1. NIH health care worker that is anticipated to be involved with the clinical care of SARS patients
   2. The ability to understand and willingness to sign a written consent form.

   A health care worker is defined as anyone involved with patient care or patient contact.

   Note: this group may be enrolled prior to SARS patients hospitalized at the clinical center.

   EXCLUSION CRITERIA:

   Probable SARS Exclusion Criteria:
   1. Age less than 18 years old.
   2. Known pregnancy or positive urine/blood pregnancy test.

   Suspected SARS Exclusion Criteria:
   1. Meets inclusion criteria for SARS
   2. Age less than 18 years old.
   3. Known pregnancy or positive urine/blood pregnancy test.

   Close Contact Exclusion Criteria:
   1. Less than 10 kg.
   2. Subjects who meet criteria for SARS or Suspected SARS

   Recovered SARS Exclusion Criteria
   1. Less than 10 kg.
   2. Temperature greater than 100.4 F (38.0 C) or symptoms of active respiratory illness

   Health Care Worker Surveillance Exclusion Criteria

   No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-11-05; Study Completion 2010-12-27

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Update: Outbreak of severe acute respiratory syndrome--worldwide, 2003. MMWR Morb Mortal Wkly Rep. 2003 Mar 28;52(12):241-6, 248. PMID 12680518
- [Background] Gilbert BE, Knight V. Biochemistry and clinical applications of ribavirin. Antimicrob Agents Chemother. 1986 Aug;30(2):201-5. doi: 10.1128/AAC.30.2.201. No abstract available. PMID 2876677
- [Background] Stein DS, Creticos CM, Jackson GG, Bernstein JM, Hayden FG, Schiff GM, Bernstein DI. Oral ribavirin treatment of influenza A and B. Antimicrob Agents Chemother. 1987 Aug;31(8):1285-7. doi: 10.1128/AAC.31.8.1285. PMID 3307623